CLINICAL TRIAL: NCT06889415
Title: The Frequency of Osteosarcopenia in Patients With Rheumatoid Arthritis and the Factors Affecting the Sarcopenia-osteoporosis Relationship
Brief Title: Rheumatoid Arthritis and Osteosarcopenia: Associated Factors
Status: Recruiting | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ilhan çağlar kaya, DOCTOR, Konya Beyhekim Training and Research Hospital
Other Study IDs: KBEAH-FTR-İK-01
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Osteosarcopenia; Rheumatoid Arthritis (RA); Sarcopenia
Keywords: osteosarcopenia; sarcopenia; Ultrasonography; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Sarcopenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rheumatoid arthritis grups: It includes females and males over the age of 50 who meet the RA diagnostic criteria according to the ACR/EULAR 2010 criteria.
  Interventions: Diagnostic Test: Osteosarcopenia in Patients with Rheumatoid Arthritis
- healty control grups: It includes females and males over the age of 50 who do not meet the exclusion criteria.
  Interventions: Diagnostic Test: Osteosarcopenia in Healthy Control Group

INTERVENTIONS:
Diagnostic Test: Osteosarcopenia in Patients with Rheumatoid Arthritis — The prevalence of osteosarcopenia will be examined in this group. Sarcopenia will be categorized into 4 groups. Both the prevalence of osteosarcopenia and the subgroups of sarcopenia will be compared with the healthy control group. Through this comparison, we will explain the relationship between sarcopenia and osteoporosis, the factors affecting this relationship, and the changes in fall and fracture risk using various questionnaires and tests.
  Groups: rheumatoid arthritis grups
Diagnostic Test: Osteosarcopenia in Healthy Control Group — The prevalence of osteosarcopenia will be examined in this group. Sarcopenia will be categorized into 4 groups. The relationship between sarcopenia and osteoporosis, the factors affecting this relationship, and the risk of falls and fractures will be evaluated using various questionnaires and tests.
  Groups: healty control grups

SUMMARY:
Our study is a cross-sectional study, and its aim is to compare and analyze the prevalence of sarcopenia and osteoporosis in patients with rheumatoid arthritis (RA) with a control group and to reveal the impact of sarcopenia on osteoporosis, fall risk, and fracture risk. This prospective cross-sectional study will include 100 rheumatoid arthritis patients and 100 healthy controls, matched for age and sex. Patients will be consecutively and meticulously enrolled based on inclusion and exclusion criteria.

A detailed medical history and examination will be performed on the patients, and their clinical and sociodemographic characteristics will be recorded. Blood tests for RA (RF, Anti-Cyclic Citrullinated Peptide (anti-CCP), CRP, ESR) and disease activity levels (DAS28) will be recorded. The prevalence of osteosarcopenia will be assessed in both the RA and healthy control groups.These groups will be evaluated using various scales and tests (including power, performance tests) including musculoskeletal ultrasonographic measurements and clinical functional assessment tests. he sarcopenic group will be categorized based on the level of sarcopenia, according to the new ISarcoPRM criteria (non-sarcopenic, dynapenic, sarcopenic, and severe sarcopenic). Osteosarcopenia will be evaluated for both groups, and the collected data will be analyzed with primary and secondary outcomes. The analysis will explore the potential relationships between rheumatoid inflammation, sarcopenia, and osteoporosis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, inflammatory joint disease that affects 5 out of 1,000 adults worldwide. The disease affects women 2 to 3 times more frequently than men and can occur at any age. The most common period for its onset is typically in the sixth decade (late 50s to 60s). In patients with rheumatoid arthritis, sarcopenia and osteopenia-osteoporosis are two commonly observed clinical conditions. Osteoporosis has been reported to be approximately twice as common in RA patients compared to the general population. The prevalence of osteoporosis in RA patients ranges from 6.3% to 36.3% in the hip region and from 12.3% to 38.9% in the spine region. Additionally, the prevalence of sarcopenia in RA patients is 21%.

Osteopenia/osteoporosis and sarcopenia are two commonly observed conditions in patients with rheumatoid arthritis (RA). Various factors increase the risk of sarcopenia in RA. These include reduced physical activity, increased levels of TNF-α and IL-1β, elevated energy expenditure at rest, increased CRP levels, and secondary immobility resulting from joint pain and stiffness.

Chronic inflammation in rheumatoid arthritis (RA) is known to increase osteoclast differentiation and suppress the osteogenesis process. In RA patients, the presence of antibodies against OPG, which inhibits RANKL, has been detected. Additionally, levels of Dickkopf-related protein 1 (DKK-1), which inhibits the Wnt signaling pathway, have been shown to be higher in the serum of RA patients compared to healthy controls. The prevalence of osteoporosis in rheumatoid arthritis patients has been reported to be more than twice that of the general population. For these reasons, the detection and prevention of osteosarcopenia in patients with rheumatoid arthritis should be considered an important comorbidity.

Sarcopenia is a syndrome characterized by the progressive and general loss of skeletal muscle mass and strength, carrying the risk of negative outcomes such as physical disability, low quality of life, and death. Although sarcopenia is typically associated with elderly individuals, it can also occur in younger individuals due to various diseases or conditions. Since its prevalence is higher in older adults compared to other age groups, it can also be referred to as a geriatric syndrome.

Various imaging methods such as computed tomography (CT), magnetic resonance imaging (MRI), dual-energy X-ray absorptiometry (DXA), bioimpedance analysis, and ultrasound can be used to determine muscle mass in the diagnosis of sarcopenia.

Osteoporosis is a systemic skeletal disease characterized by a decrease in bone mass and a deterioration of the structural integrity of bone tissue, which increases bone fragility and creates a risk of fractures. The World Health Organization (WHO) defines osteoporosis through measurements made using dual-energy X-ray absorptiometry (DXA). According to this definition, the T-score in the lumbar spine, femoral neck, or distal third of the radius is evaluated as follows: T-score ≥ -1.0 is normal, between -1.0 and -2.5 is osteopenia, and T-score ≤ -2.5 is considered osteoporosis. Additionally, if the T-score is below -2.5 and one or more osteoporotic fractures are present, this condition is referred to as established osteoporosis.

Sarcopenia is evaluated based on specific criteria. Although the information may change over time, it is important to consider muscle strength, muscle mass, and physical performance when diagnosing sarcopenia today.

Recently, the STAR study has been published, emphasizing the importance of regional muscle mass measurements in the diagnosis of sarcopenia. The study showed that the thickness of the anterior thigh muscle is the parameter that decreases the most with aging, and this measurement has a stronger correlation with height and BMI. In this regard, it is recommended to use the STAR value, obtained by dividing the anterior thigh muscle thickness measured by ultrasound by BMI, in the diagnosis of sarcopenia. The STAR threshold value has been set as <1.0 for women and <1.4 for men.

The formula is:

STAR = Anterior thigh muscle thickness (mm) / Body Mass Index (BMI) (kg/m²)

International Society of Physical and Rehabilitation Medicine, ISPRM (2021) has published a new sarcopenia diagnostic algorithm, which also includes the STAR study and ISarcoPRM recommends screening for all older adults and adults with RAS-associated disorders.

ISarcoPRM has set cut-off values of ≥12 seconds for the sit-to-stand test and <32 kg for grip strength in men and <19 kg in women to identify low muscle function. Initially, both tests are recommended. If low values are detected in either of these tests, the patient is considered to have "probable sarcopenia."

In individuals diagnosed with probable sarcopenia, it is recommended to measure the anterior thigh muscle thickness using ultrasound and calculate the STAR value. If the STAR value is below the threshold level determined by gender, the individual is classified as having "sarcopenia." Additionally, if the walking speed is ≤ 0.8 m/s and/or the individual cannot rise from a chair without support, this condition is defined as "severe sarcopenia."

If at least one of the patient's muscle function tests is low but the STAR value is normal, the patient is considered to have "dynapenia.

In our study, in addition to anterior thigh thickness, Achilles tendon thickness will also be measured. There is insufficient research explaining the relationship between Achilles tendon thickness and sarcopenia or osteoporosis. In this study, we will also investigate whether there is a relationship between Achilles tendon thickness and sarcopenia and/or osteoporosis.

There are few studies examining the relationship between RA, osteoporosis, and sarcopenia with heterogeneous methodologie. Therefore, the aim of this study is to evaluate the prevalence of osteosarcopenia in RA patients and control groups, and to investigate the impact of sarcopenia, along with the effects of inflammation, on osteoporosis, fall, and fracture risk. By evaluating sarcopenia according to the ISarcoPRM criteria, the study aims to address the gap in the literature with a unique and robust original methodologies.

ELIGIBILITY:
Inclusion criteria:

1. Being diagnosed with RA according to the ACR/EULAR 2010 criteria
2. Being a female or male over the age of 50
3. Having the mental and physical capacity to complete the study questionnaires and tests
4. Providing voluntary consent to participate in the study by signing the Informed Consent Form

Exclusion Criteria:

1. Having an acute illness/disability or significant cognitive impairment that prevents understanding and performing the required tests
2. Having thyroid or parathyroid disease, uncontrolled diabetes, Cushing's syndrome, anemia.
3. History of malignancy
4. Severe cardiovascular disease, enal failure, advanced-stage COPD, decompensated liver disease
5. History of gastrointestinal (GIS) surgery

7-Having another coexisting autoimmune/inflammatory rheumatic disease (e.g., SLE, Ankylosing Spondylitis, etc.), psoriatic arthritis, vasculitis, familial Mediterranean fever...)

8-Having severe/symptomatic hand osteoarthritis and/or deformities

9-Severe/symptomatic osteoarthritis in the knee, lumbar, hip, or ankle region

10-Having Carpal Tunnel Syndrome, De Quervain, lateral epicondylitis, cubital tunnel syndrome or a history of traumatic hand injury

11-Having a significant neurological disease, stroke, MS, myopathy, Parkinson's disease, radiculopathy/polyneuropathy/brachial plexopathy or others nerve root compressions

12-History of surgical intervention on the upper and lower extremities or spine

13-Having severe kyphosis or scoliosis

14-Having any others disease causing balance disorders (neurological, orthopedic, metabolic, etc.)

15-Having a major/significant psychiatric disorder (based on the medical history, and hospital records)

16-Current use of androgens or estrogens

17-Having prostheses, being fully dependent, or immobilized

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include consecutively 100 patients with RA aged 50 and over, who have been diagnosed according to the ACR/EULAR 2010 classification criteria (who have visited the Physical Medicine and Rehabilitation and Rheumatology outpatient clinics) and 100 age- and gender-matched healthy control subjects.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia assessment | baseline
  According to the ISarcoPRM (2021) diagnostic algorithm and the reference values based on its threshold, participants were categorized into sarcopenia groups (no sarcopenia, dynapenia, sarcopenia, severe sarcopenia).
Osteoporosis assessment/dual-energy X-ray absorptiometry | baseline
  Dual-energy X-ray absorptiometry (DXA) measurements will be reviewed. In the lumbar spine, femoral neck, or total femur; a T score ≥ -1.0 is considered normal, -1 > T score > -2.5 is osteopenia, and T score ≤ -2.5 is defined as osteoporosis.
Balance and Gait Assessment Scale | baseline
  This scale is an important tool to evaluate the individual's functional status and daily living activities. The scale consists of a maximum of 16 points for balance and a maximum of 12 points for walking, for a total of 28 points. Individuals who score 26 or below on the scale are thought to have a problem; For those with scores of 19 or below, it is observed that the risk of self-falling increases fivefold compared to normal individuals.

SECONDARY OUTCOMES:
Fracture Risk Assessment Tool (FRAX) | baseline
  The Fracture Risk Assessment Tool (FRAX) will be calculated using the Turkish population version. The World Health Organization developed this web-based scoring system to assess the 10-year risk of hip fractures or major osteoporotic fractures based on fracture risk factors. According to the FRAX scoring system, treatment is recommended when the major osteoporotic fracture risk is 20% or higher, and the 10-year hip fracture risk is 3% or above.
Health Assessment Questionnaire, HAQ | baseline
  It can assess RA patients in all dimensions, such as disability and discomfort. It includes sections that evaluate disability with 20 questions, pain with one question, and global health status with one question. The disability index includes 8 areas that assess dressing and self-care, getting up, eating, walking, hygiene, reaching, grasping, and normal daily activities. Each section is scored individually, and the average of the 8 sections is recorded. This survey score ranges from 0 to 3. As the score increases, the health condition worsens.
Handgrip Strength Test | baseline
  According to the protocol recommended by the American Society of Hand Therapists in 1992, measurements will be taken while patients are seated, with the shoulder in neutral rotation and adduction, the elbow at 90° flexion, the forearm in a neutral position, and the wrist in 30 degrees of dorsiflexion. Patients will be instructed to squeeze the dynamometer with all their strength using similar words and tone. Grip strength will be measured for both hands. Measurements will be taken three times with 1-minute rest intervals, and the maximum value will be recorded. According to the ISarcoPRM (2021) diagnostic algorithm, values below <32 kg for men and <19 kg for women will be considered as reduced muscle strength.
chair rise test | baseline
  The five-time chair rise test is a measure used to assess lower extremity muscle strength. The patient will be asked to cross their arms over their chest and sit down and stand up from the chair five times as quickly as possible, with the time being recorded. If the time exceeds 12 seconds, it will be considered a reduction in muscle strength.
Anterior Thigh Muscle Thickness Measurement | baseline
  Participants will be evaluated while lying in a supine position, with their arms and legs extended and muscles relaxed. The measurement region will be selected as the midpoint between the anterior superior iliac spine and the upper pole of the patella. The ultrasound probe will be positioned in the axial plane at a 90-degree angle to the muscle extension. During imaging, measurements will be taken with a generous amount of gel applied, without any compression. The anterior thigh muscle thickness will be determined as the total thickness of the rectus femoris and vastus intermedius muscles, and the distance between the outer fascia of the rectus femoris and the femur periosteum will be used as the reference. Measurements will be repeated three times, and the average value will be recorded in mm. The noted muscle thickness will be divided by the participant's BMI to calculate the STAR value.
6-meter Walking Test | baseline
  The patient will be asked to walk a 6-meter distance at their normal walking speed, as in daily life. The time taken to complete the 6 meters will be recorded in seconds. The 6-meter walking speed will be calculated in meters per second (m/s), and speeds below 0.8 m/s will be considered as low walking speed.
Achilles tendon thickness measurement | baseline
  There is insufficient research explaining the relationship between Achilles tendon thickness and sarcopenia and osteoporosis. In this study, we will also examine whether there is a relationship between Achilles tendon thickness and sarcopenia and/or osteoporosis.
  Participants will lie in a prone position with their feet hanging off the examination table. The tendon thickness will be measured axially (at the thickest point between the epitenons) at the level of the lateral malleolus.
VAS pain (pain intensity) | baseline
  A horizontal visual analog scale (VAS) will be used to assess the participants' pain levels. A 10 cm long line will be drawn on a blank paper, with the left end marked as "0" (no pain) and the right end marked as "10" (unbearable pain). Participants will be asked to indicate the intensity of their pain by marking an appropriate point on this line.

CONTACTS AND LOCATIONS:
Overall Officials: İlhan ç KAYA, Principal Investigator — Konya Beyhekim Training and Research Hospital Physical Medicine and Rehabilitation Clinic
Locations (1):
- Konya Beyhekim Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucukdeveci AA, Sahin H, Ataman S, Griffiths B, Tennant A. Issues in cross-cultural validity: example from the adaptation, reliability, and validity testing of a Turkish version of the Stanford Health Assessment Questionnaire. Arthritis Rheum. 2004 Feb 15;51(1):14-9. doi: 10.1002/art.20091. PMID 14872450
- [Background] Çifçili S, Ünalan PC. Yaşlılarda fonksiyonel kayıplara yaklaşım. Turkish Journal of Family Practice. 2004;8(4):166-73
- [Background] Ozcakar L, Kara M, Chang KV, Bayram Carli A, Hung CY, Tok F, Wu CH, Akkaya N, Hsiao MY, Tekin L, Wang TG, Ulasli AM, Chen WS, De Muynck M. EURO-MUSCULUS/USPRM. Basic Scanning Protocols for Ankle and foot. Eur J Phys Rehabil Med. 2015 Oct;51(5):647-53. Epub 2015 Sep 8. PMID 26351106
- [Background] Chiu YH, Liao CL, Chien YH, Wu CH, Ozcakar L. Sonographic evaluations of the skeletal muscles in patients with Pompe disease. Eur J Paediatr Neurol. 2023 Jan;42:22-27. doi: 10.1016/j.ejpn.2022.12.002. Epub 2022 Dec 6. PMID 36508847
- [Background] van Riel PL, Renskers L. The Disease Activity Score (DAS) and the Disease Activity Score using 28 joint counts (DAS28) in the management of rheumatoid arthritis. Clin Exp Rheumatol. 2016 Sep-Oct;34(5 Suppl 101):S40-S44. Epub 2016 Oct 18. PMID 27762189
- [Background] Pinheiro PA, Passos TD, Coqueiro Rda S, Fernandes MH, Barbosa AR. [Motor performance of the elderly in northeast Brazil: differences with age and sex]. Rev Esc Enferm USP. 2013 Feb;47(1):128-36. doi: 10.1590/s0080-62342013000100016. Portuguese. PMID 23515812
- [Background] Maggio M, Ceda GP, Ticinesi A, De Vita F, Gelmini G, Costantino C, Meschi T, Kressig RW, Cesari M, Fabi M, Lauretani F. Instrumental and Non-Instrumental Evaluation of 4-Meter Walking Speed in Older Individuals. PLoS One. 2016 Apr 14;11(4):e0153583. doi: 10.1371/journal.pone.0153583. eCollection 2016. PMID 27077744
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Adami G, Saag KG. Osteoporosis Pathophysiology, Epidemiology, and Screening in Rheumatoid Arthritis. Curr Rheumatol Rep. 2019 May 23;21(7):34. doi: 10.1007/s11926-019-0836-7. PMID 31123839
- [Background] Torii M, Hashimoto M, Hanai A, Fujii T, Furu M, Ito H, Uozumi R, Hamaguchi M, Terao C, Yamamoto W, Uda M, Nin K, Morita S, Arai H, Mimori T. Prevalence and factors associated with sarcopenia in patients with rheumatoid arthritis. Mod Rheumatol. 2019 Jul;29(4):589-595. doi: 10.1080/14397595.2018.1510565. Epub 2018 Sep 11. PMID 30092163
- [Background] Kanis JA. Diagnosis of osteoporosis and assessment of fracture risk. Lancet. 2002 Jun 1;359(9321):1929-36. doi: 10.1016/S0140-6736(02)08761-5. PMID 12057569
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Barone M, Viggiani MT, Anelli MG, Fanizzi R, Lorusso O, Lopalco G, Cantarini L, Di Leo A, Lapadula G, Iannone F. Sarcopenia in Patients with Rheumatic Diseases: Prevalence and Associated Risk Factors. J Clin Med. 2018 Dec 1;7(12):504. doi: 10.3390/jcm7120504. PMID 30513782
- [Background] Haugeberg G, Uhlig T, Falch JA, Halse JI, Kvien TK. Bone mineral density and frequency of osteoporosis in female patients with rheumatoid arthritis: results from 394 patients in the Oslo County Rheumatoid Arthritis register. Arthritis Rheum. 2000 Mar;43(3):522-30. doi: 10.1002/1529-0131(200003)43:33.0.CO;2-Y. PMID 10728744
- [Background] Aletaha D, Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018 Oct 2;320(13):1360-1372. doi: 10.1001/jama.2018.13103. PMID 30285183